CLINICAL TRIAL: NCT05397925
Title: Effectiveness of a Training Program for Self-management of the Substance Addiction Consequences - Protocol for a Randomized Controlled Trial
Brief Title: Effectiveness of a Training Program for Self-management of the Substance Addiction Consequences - a Study Protocol
Acronym: ADSProgram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nursing School of Lisbon (Other)
Collaborators: Center for Health Technology and Services Research (Other)
Responsible Party: Principal Investigator, Paulo Rosário Carvalho Seabra, Prof., Nursing School of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6649/CES/2020
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Substance Related Disorders
Keywords: Substance Related Disorder; Nursing Interventions; self management; training program; opiate substitution treatment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: ADSProgram - Program for self-management of Substance Dependence. It is a program based on a holistic view of the person and the ability to help people to reach their full potential based on their personal resources. It is also based on the need to focus interventions on the assessment and monitoring of substance addiction consequences. Is a harm reduction paradigm program to support self-management of this chronic condition. Aim: Training for self-management of substance addiction consequences; Promote adherence to the therapeutic project; Promote positive mental health. Therapeutic strategies - The principles of motivational interviewing, brief interventions with cognitive behavioral orientation and based on the assumptions of "helping relationship" to support the process of change.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Eligible participants will be recruited by the nurses of each institution. A baseline assessment will be carried out and the instruments will be applied after informed consent by participants. Participants will be randomly allocated to ADSProgram (experimental group). The control group will receive the treatment as usual (TAU). In both groups will be maintained the TAU. All participants will be re-assessed at the end of the program by assistant researchers. Principal Investigator will receive documental anonymized data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADSProgram (Experimental): This is the experimental arm of the study. This includes receiving the novel/experimental ADSProgram. Therapy description withheld to protect the integrity of the study.
  Intervention: ADSprogram
  Interventions: Behavioral: ADSProgram - Self management for substance dependence program
- Treatment as usual (Active Comparator): This is the control arm of the study. This includes receiving the standard of care on nursing Consultations on a medication-based program and multidisciplinary regular care. Therapy description withheld to protect the integrity of the study.
  Intervention: Nursing Consultation
  Interventions: Behavioral: Treatment as usual - Regular nursing consultation on a medication-based program

INTERVENTIONS:
Behavioral: ADSProgram - Self management for substance dependence program — GENERAL STRUCTURE OF THE MODEL - 8 sessions: One initial - assessment; 1 to 6 Intermediates - empowerment (Flexible number of intermediate sessions according to the person's need and accessibility, interlude 1 week minimum, up to a maximum of 3 weeks); 1 Final - autonomy; Duration of sessions: 20-60 min; Context: Outpatient specialized addictions unit. Private room needed; Preferred approach: Individual, face-to-face or virtual consultation. Complementary approach: In groups of up to 4 people, when peer support or sharing feelings are needed: Clinical focus 1 - Concerning the problematic use of substances, 2 - Related to health knowledge in general, 3 - Related to health-seeking behavior and adherence, 4 - Related to self-knowledge and well-being, 5 - Related to social role and personal dignity, 6 - Related to the family process.
  Arms: ADSProgram
Behavioral: Treatment as usual - Regular nursing consultation on a medication-based program — Regular individual assessment on: substance used (kind of substance, consumption way, frequency), way of living, social relationship, health status nursing diagnoses. To support on this, therapeutic interventions, medication delivery and management support.
  Arms: Treatment as usual

SUMMARY:
The substance dependent population has many health needs in which it is necessary to invest in competent approaches with more evidence. The main needs can be minimized when people are trained for self-care (abstinence, risk reduction and harm minimization) and for the necessary adaptations to the impact that these addictive behaviors and dependencies have on their lives and their families' lives.

Nursing can play a leading role in interventions aimed at reducing stigma and self-stigma, increasing users' knowledge for recovery, responding to the needs of older consumers, and helping training for self-management of substance dependence. However, about "nursing intervention programs" with people dependent on substances, the evidence is scarce. In many chronic illness situations, people need programs to train and develop a better capacity for self-management of their health situation.

Nurses in the Addictive Behaviors area globally closely linked to medication-based programs, hold consultations, manage programs and there is evidence of results that are sensitive to nursing care, however, professionals can and should seek new systematic approaches in response to people's needs and should seek to increase the level of evidence of the result of the interventions.

This complex phenomenon can be accompanied by the ability of individuals to manage the severity of the consequences. Based on all this, the following research question emerge: How effective could be an intervention program for training people to manage substance addiction consequences?

A randomized controlled trial that will be realized in one specialized unit on addictions, in Lisbon area. Pilot study will be carried out initially. The total sample will be constituted by individuals with substance use disorders, in a medication-based outpatient program, that will be receiving the ADSProgram (experimental group (n=30) and control group receiving treatment as usual (n=30). Both will be aplied for 21 weeks maximum.

The General Objective for this research is "To evaluate the effectiveness of a training program for self-management of the substance addiction consequences, with people integrated in medication-based programs".

The hypotheses to be tested is that this program is effective to reduce substance addiction consequences.

DETAILED DESCRIPTION:
The substance dependent population has many health needs in which it is necessary to invest in competent approaches, with more evidence. The main needs can be minimized when people are trained for self-care (abstinence, risk reduction and harm minimization) and for the necessary adaptations to the impact that these addictive behaviors and dependencies have on their lives and their families' lives. It should be noted that people with addictive behavior, who have health needs, call for a more active role for nurses in their follow-up processes, value respect for care and value their co-decision on the care plan.

Nursing can play a leading role in interventions aimed to reduce stigma and self-stigma, increasing users' knowledge for recovery, responding to the needs of older consumers, and help to train for self-management of substance dependence. However, about "nursing intervention programs" with people dependent on substances, the evidence is scarce. In many chronic illness situations, people need programs to train and develop a better capacity for self-management of their health situation.

Nurses in the Addictive Behaviors area globally closely linked to medication-based programs, hold consultations, manage programs and there is evidence of results that are sensitive to nursing care, however, professionals can and should seek new systematic approaches in response to people's needs and should seek to increase the level of evidence of the outcomes of the interventions.

This complex phenomenon can be accompanied by the ability of individuals to manage the severity of the consequences, for which there are instruments to assess, and to improve "positive mental health" aimed to deepening persons state of health and changes that occur over time. Positive Mental Health can be defined as a value in itself (feeling good), a way of interpreting the environment in which participants find themselves to adapt and carry out changes that allow this adaptation. Mental health can be seen as an indicator of integration and adaptation and is often impaired by substance use.

Based on all this, the following research question emerge: How effective could be an intervention program for training people to manage substance addiction consequences?

The General Objective for this research is "To evaluate the effectiveness of a training program for self-management of the substance addiction consequences, with people integrated in medication-based programs".

The hypotheses to be tested is that this program is effective to reduce substance addiction consequences.

Based on these assumptions, investigators intend to carry out, a pilot (first) and a rondomized control study following the methodological recommendations for the development of complex interventions by the Medical Research Council - FEASIBILITY AND PILOTING - Testing, application and evaluation - Pilot study with the implementation of the training program for self-management of substance addiction consequences and ASSESSMENT (Randomized controlled experimental study).

A randomized controlled trial that will be realized in one specialized unit on addictions, in Lisbon area. Pilot study will be carried out initially with individuals with substance use disorders, in a medication-based outpatient program, that will be receiving the ADSProgram (experimental group (n=15) and control group receiving treatment as usual (n=15). In experimental group the ADSProgram will be applied for 21 weeks maximum for each patient. After pilot study research team intend to perform the RCT with experimental group (n=30) and control group (n=30) also.

From the day on which the selection of participants begins, participants will be randomly invited to participate in the study, starting with the first user evaluated in consultation after checking their criterion value on the substance addiction consequences scale (<=48). Some participants will be evaluated during the chronological course of the regular medication-based program, assisted in the nursing consultations and by the remaining professionals (control group). Others (with the same regular interventions) will be cumulatively invited to participate in the study, integrating the sample that will receive the interventions of the program (experimental group). Randomization will be done by previous determination of selected numbers by an online randomization application. Two sets of numbers will be created - the first set to control group and the second set to experimental group. Sample numbers will be created because when someone refuses to participate, nurses will select the next number in the randomized sets to different study arms. The enrollment will be strict since the first one in consultation and for those who accept to participate.

Also the sample will be theoretical randomized in face the homogenous comparative sample (sex, age groups, type of medication program and length on the program).

When completing the sample of 15 participants in the control group and 15 in the experimental group, the data will be analyzed comparing the effect between groups in reducing the substance addiction consequences. The size of the dropouts and their extension will also be analyzed in relation to the variables established for the homogeneity of the samples. After this evaluation of the results of the pilot study, the selection of participants will proceed until 30+30, with the initial sample being able to integrate the final study if the parallel sample remains with similar characteristics.

Descriptive, inferential, and multivariable statistical analyses will be used to describe participants, determine the effect size change and to determine which variables are related to better or worst severity. Missing data will be managed case by case due to the different variables under study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Included in a medication-based program for at least 5 weeks in a specialized unit
* Accept to be followed in a nursing consultation.
* Severe severity (=<48 on Substance addiction Consequences (SAC) scale

Exclusion Criteria:

* Patients with impairment of thinking and perception
* Aggressive behaviour
* Psychomotor agitation.
* Patient with severe cognitive impairment (<17 on Montreal Cognitive Assessment (MoCA))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Substance Addiction Consequences Scale | Up to 21 weeks
  It has 16 items, with a 5-point Likert scale (1-5), between severe and none, the higher the value, the lower the severity. The possible response range is between 16 and 80, with the value 48 referring to 50% of the possible range. Made up of four dimensions (psychological and family factors, physical and cognitive factors, economic and labor factors and self-care factors). The average of each item can be obtained in the range 1-5, with the midpoint 2.5. In each dimension, investigators calculate the average adjusted to the number of items.
Positive Mental Health Questionary | Up to 21 weeks
  The questionnaire contains a series of statements about the way of thinking, feeling and acting, presenting 39 questions grouped into six dimensions (personal satisfaction; prosocial attitude; self-control; autonomy; problem-solving ability and personal fulfillment; interpersonal relationship skills). Is rated on a Likert scale from 1 to 4 points, with the following response possibilities: always or almost always (1 point), most of the time (2 points), sometimes (3 points) ), rarely or never (4 points). Higher the value, better the Positive Mental Health (PMH).

SECONDARY OUTCOMES:
Sections attendance rate | Up to 21 weeks
  (Number of attendance/Number of programed sections) x 100
Nursing diagnoses status improvement | Up to 21 weeks
  (Number of participants who improve the status on half of diagnoses/Total sample who finalized the program) x 100

OTHER OUTCOMES:
Sex of paticipants | Baseline
  sex
Age of participants | Baseline
  Age group
Type of the program | Baseline
  Type of medication program
Lengh of medication program | Baseline
  lengh on the program

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Seabra, Principal Investigator — Nursing School of Lisbon
Locations (2):
- Portugal (2):
  - ETET Barreiro, Barreiro
  - Setubal Peninsula Integrated Response Center - THE REGIONAL HEALTH ADMINISTRATION OF LISBON AND VALE DO TEJO, Barreiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seabra PRC, Amendoeira JJP, Sa LO, Capelas MLV. Clinical Validation of the Portuguese Version of "Substance Addiction Consequences" Derived from the Nursing Outcomes Classification. Issues Ment Health Nurs. 2018 Sep;39(9):779-785. doi: 10.1080/01612840.2018.1462870. Epub 2018 Aug 15. PMID 30111209
- [Background] Seabra P, Brantes AL, Sequeira R, Sequeira A, Nunes I, Sequeira C. Aceitabilidade e aplicabilidade de um programa de intervenção com usuários dependentes de substâncias. Submitted. 2021;
- [Background] Sequeira C, Carvalho JC, Sampaio F, Sá L, Lluch-Canut T, Roldán-Merino J. Avaliação das propriedades psicométricas do Questionário de Saúde Mental Positiva em estudantes portugueses do ensino superior. Rev Port Enferm Saúde Ment. 2014;(11):45-53.
- [Background] van Schie D, Castelein S, van der Bijl J, Meijburg R, Stringer B, van Meijel B. Systematic review of self-management in patients with schizophrenia: psychometric assessment of tools, levels of self-management and associated factors. J Adv Nurs. 2016 Nov;72(11):2598-2611. doi: 10.1111/jan.13023. Epub 2016 Jun 13. PMID 27200500
- [Background] Van de Velde D, De Zutter F, Satink T, Costa U, Janquart S, Senn D, De Vriendt P. Delineating the concept of self-management in chronic conditions: a concept analysis. BMJ Open. 2019 Jul 16;9(7):e027775. doi: 10.1136/bmjopen-2018-027775. PMID 31315862
- [Result] Sampaio FM, Sequeira C, Lluch Canut T. Content Validity of a Psychotherapeutic Intervention Model in Nursing: A Modified e-Delphi Study. Arch Psychiatr Nurs. 2017 Apr;31(2):147-156. doi: 10.1016/j.apnu.2016.09.007. Epub 2016 Sep 14. PMID 28359426